CLINICAL TRIAL: NCT03289741
Title: A Pilot Study To Evaluate Patient Experience With the Somatostatin Analogs Octreotide Long Acting Release and Lanreotide During the Treatment of Advanced, Nonfunctional, Well Differentiated Neuroendocrine Tumors
Brief Title: A Study to Evaluate Patient Experience in the Therapy of Neuroendocrine Tumors Treated With Octreotide Long Acting Release Versus Lanreotide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-422
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors
Keywords: Octreotide; Lanreotide; 17-422
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Octreotide; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Two-arm randomized design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Octreotide then Lanreotide (Experimental): Each patient on study will receive three injections of intramuscular (IM) octreotide Long Acting Release (LAR). Octreotide LAR for 3 injections followed by lanreotide for 3 injections
  Interventions: Drug: Octreotide; Drug: LAR Lanreotide; Behavioral: Questionnaires
- Lanreotide then Octreotide (Experimental): Each patient on study will receive three injections of deep subcutaneous (subq) lanreotide. Lanreotide for 3 injections followed by octreotide LAR for 3 injections
  Interventions: Drug: Octreotide; Drug: LAR Lanreotide; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Octreotide — Patients will receive three monthly injections every 28 (+/- 3) days. Octreotide LAR for 3 injections followed by lanreotide for 3 injections
Drug: LAR Lanreotide — Patients will receive three monthly injections every 28 (+/- 3) days. Lanreotide for 3 injections followed by octreotide LAR for 3 injections
Behavioral: Questionnaires — Baseline questionnaire, Post-treatment questionnaire (after the first 3 injections), Preference questionnaire and Pain Score Diary.

SUMMARY:
This study is being done to evaluate differences in patient experience during treatment with octreotide LAR and lanreotide.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial
* ≥ 18 years of age
* Histologically- or cytologically- confirmed locally advanced or metastatic WDNET
* SSA therapy is recommended by physician for disease management, and has not yet begun
* ECOG performance status of 0, 1, or 2

Exclusion Criteria:

* Currently participating in a study of an investigational agent
* Prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent

  *Note: Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study
* No concurrent chemotherapy or targeted small molecule therapy
* If received major surgery, not recovered adequately from the toxicity and/or complications from the intervention prior to starting the study
* Known additional malignancy that is progressing or requires active treatment
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Raj, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Result] Raj N, Cruz E, O'Shaughnessy S, Calderon C, Chou JF, Capanu M, Heffernan O, DeMore A, Punn S, Le T, Hauser H, Saltz L, Reidy-Lagunes D. A Randomized Trial Evaluating Patient Experience and Preference Between Octreotide Long-Acting Release and Lanreotide for Treatment of Well-Differentiated Neuroendocrine Tumors. JCO Oncol Pract. 2022 Sep;18(9):e1533-e1541. doi: 10.1200/OP.22.00055. Epub 2022 Jun 20. PMID 35724357
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octreotide Then Lanreotide | Lanreotide Then Octreotide
Started | 26 | 25
Completed | 22 | 22
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide Then Lanreotide | Lanreotide Then Octreotide | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Full Range); unit: years] | 63 [40 to 83] | 67 [47 to 87] | 65 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 21 | 19 | 40
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Scores at 3 Months
Description: Patients will rate, on a numeric scale of 0 to 10, with 0 being No pain" to 10 being "Worst pain ever" the pain or discomfort experienced with the SSA injection.
Time Frame: 3 months
Population: The mean pain scores for each treatment arm is appropriately reported below.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Octreotide Then Lanreotide | Lanreotide Then Octreotide
Number analyzed (Participants) | 26 | 25
scores on a scale
  Octreotide, first intervention (3 months): number analyzed (Participants) | 26 | 0
  Octreotide, first intervention (3 months) | 2.4 [0 to 10] |
  Lanreotide, second intervention (6 months): number analyzed (Participants) | 26 | 0
  Lanreotide, second intervention (6 months) | 2.4 [0 to 10] |
  Lanreotide, first intervention (3 months): number analyzed (Participants) | 0 | 25
  Lanreotide, first intervention (3 months) |  | 1.9 [0 to 10]
  Octreotide, second intervention (6 months): number analyzed (Participants) | 0 | 25
  Octreotide, second intervention (6 months) |  | 1.9 [0 to 10]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Groups:
- Octreotide: Each patient on study will receive three injections of intramuscular (IM) octreotide Long Acting Release (LAR). Octreotide LAR for 3 injections followed by lanreotide for 3 injections. Participants are assigned to one arm of the study and they remain on that arm for the duration of the study.
  Octreotide: Patients will receive three monthly injections every 28 (+/- 3) days. Octreotide LAR for 3 injections followed by lanreotide for 3 injections
  LAR Lanreotide: Patients will receive three monthly injections every 28 (+/- 3) days. Lanreotide for 3 injections followed by octreotide LAR for 3 injections
  Questionnaires: Baseline questionnaire, Post-treatment questionnaire (after the first 3 injections), Preference questionnaire and Pain Score Diary.
- Lanreotide: Each patient on study will receive three injections of deep subcutaneous (subq) lanreotide. Lanreotide for 3 injections followed by octreotide LAR for 3 injections. Participants are assigned to one arm of the study and they remain on that arm for the duration of the study.
  Octreotide: Patients will receive three monthly injections every 28 (+/- 3) days. Octreotide LAR for 3 injections followed by lanreotide for 3 injections
  LAR Lanreotide: Patients will receive three monthly injections every 28 (+/- 3) days. Lanreotide for 3 injections followed by octreotide LAR for 3 injections
  Questionnaires: Baseline questionnaire, Post-treatment questionnaire (after the first 3 injections), Preference questionnaire and Pain Score Diary.
Arm/Group | Octreotide | Lanreotide
All-Cause Mortality (participants affected / at risk) | 13/51 | 8/51
Serious Adverse Events (participants affected / at risk) | 13/51 | 8/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide (N=51) | Lanreotide (N=51)
Death NOS (General disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03289741/Prot_SAP_000.pdf